CLINICAL TRIAL: NCT01357785
Title: Periodontal Tissue Regeneration Using Autologous Periodontal Ligament Stem Cells: Randomized Controlled Clinical Trial
Brief Title: Periodontal Tissue Regeneration Using Autologous Periodontal Ligament Stem Cells
Acronym: PDLSC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Fa-Ming Chen, Fourth Military Medical University, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Periodontal Pocket
Keywords: Periodontal ligament stem cells; Periodontal regeneration; Clinical trial; Deep intraosseous defects
MeSH Terms: conditions — Periodontal Pocket | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cell therapy — The use of periodontal ligament stem cells for periodontal regeneration

SUMMARY:
The purpose of this clinical trial is to both clarify the efficiency of autologous periodontal ligament (PDL) stem cells to regenerate periodontal tissue in periodontitis patients with deep intraosseous defects (>5 mm) and to confirm the safety of using autologous stem cells in clinical periodontal regenerative medicine. This is a single-centre, randomized, placebo-controlled study. This study has been approved by the ethical committees of School of Stomatology, Fourth Military Medical University. The study will be conducted according to the Declaration of Helsinki.

DETAILED DESCRIPTION:
Periodontitis is an inflammatory disease that causes pathological alterations in the tooth-supporting tissues, potentially leading to tooth loss. National surveys have shown that the majority of adults in the population suffer from moderate periodontitis, with up to 15% of the population being affected by severe generalized periodontitis at some stage in their lives. The significant burden of periodontal disease and its impact on general health and patient quality of life point to the clinical need for effective management of this condition. The ultimate goal of periodontal therapy is predictably regeneration of a functional attachment apparatus destroyed by peridontitis, which involves the formation of a new cementum, periodontal ligament (PDL), and alveolar bone. To date, several therapeutic procedures have been attempted to achieve this ambitious purpose, including root surface conditioning, bone graft placement, guided tissue regeneration (GTR) and the use of enamel matrix-derived proteins or growth factors. However, current regenerative techniques that are used either alone or in combination have limitations in attaining complete and predicable regeneration, especially in advanced periodontal defects, where deep intraosseous defects have been shown to be high-risk sites for progression of periodontitis.

According to histologic evidence, the GTR technique combined with bone graft is the most predictable regenerative procedure in the treatment of such periodontal defects, although basically, current available GTR-based therapies are still crude and of poor clinical predictability. During periodontal regenerative procedures, the remaining healthy periodontal ligament (PDL) plays a key role in the regeneration of new compartments, and the cells of PDL tissues are the only cells that seem to have the capacity to form new attachment apparatus.. The regenerative capacity of the PDL itself is attributed to a few progenitor cells maintaining their proliferation and differentiation potential in the periodontium. Recent advances in stem cell biology and regenerative medicine have presented opportunities for tissue engineering in periodontal therapy. To date, a large number of studies have reported that stem cells, in conjunction with different physical matrices and growth factors, have the capacity to regenerate periodontal tissues in vivo.

It has been demonstrated that PDL-derived progenitors are committed to several developmental lineages, i.e., osteoblastic, fibroblastic and cementoblastic. This property determines the PDL cells as a desirable cell population capable of regenerating a functional periodontal attachment apparatus. It has been shown that PDL cells may prevent ankylosis and root resorption and may possibly also produce a new PDL inserted into the tooth and adjacent bone. Moreover, roots covered with alveolar bone cells induce a cementum-like tissue formation, suggesting that cementoblast and osteoblast precursors commonly originate from the alveolar bone. Thus, PDL-derived cell sources are one of the most promising candidates for cell-based therapies and tissue-engineering-associated periodontal regeneration, and positive pre-clinical results have already been achieved both in vitro and in vivo. Taken together, the results of these investigations demonstrate that PDL cells are capable of preventing epithelial down-growth and root resorption, with the periodontal healing pattern being characterized by connective tissue adaptation involving parallel bundles resting on root dentin. The formation of new bone and cementum varies from a complete absence to coverage of parts of the debrided root surfaces mainly at the borders of the defects, to a thin layer of newly formed cementum with complete new bone formation covering the entire previously denuded root surface. The heterogeneity of results obtained may be explained by the small number of specimens used, the different types of periodontal defects observed and the stability of the carriers utilized to deliver the cells (i.e., hyaluronic acid and blood clots). In addition, one may speculate that PDL cell differentiation is highly sensitive to differences in the microenvironment, resulting in different types of periodontal healing. However, the clinical application of autologous PDL-derived cells are currently lacking.

All over the world, periodontitis remains highly prevalent, can lead loss of the affected teeth, and thus threaten quality of life for middle-aged population as far as oral functions are concerned. Unfortunately in clinic, no current periodontal treatments can, at best, heal the scar in the affected region and ever regenerate lost periodontal tissue or normal structure and functionality. Considering that the "mouth" and "teeth" have various aesthetic and functional roles to play, establishing a brand-new treatment that enables the regeneration of periodontal tissue is very important. It is clear that there is both a clinical need for such treatments and a vast patient resource. Interestingly, there is mounting data that demonstrates the induction of periodontal tissue regeneration by PDL stem cells in animal models. In particular, a number of studies show that topical administration of PDL stem cells enhances periodontal tissue regeneration in models of artificial loss of periodontal tissue in beagles and non-human primates. This suggests that PDL stem cells may be safe and effective in the regeneration of periodontal tissues in periodontitis patients.

In the phase I clinical trial for 20 healthy male volunteers by local administration of autologous PDL stem cells, neither adverse reactions nor rise of any antibody were observed (unpublished data). Importantly, several groups have commenced small-scale pilot/feasibility studies, leading sufficient information to move cell-based therapy into the clinical arena. It is therefore we established this clinical protocol to further test the efficiency and safety of stem cells in the treatment of periodontal deep intraosseous defects.

ELIGIBILITY:
Inclusion Criteria:

1. Those diagnosed as having, from radiography and other results, 2- or 3-walled vertical intrabony defect 3 mm deep from the top of the remaining alveolar bone
2. Those who have accomplished initial preparation and have been showing good compliance
3. Those with mobility of the tooth to investigate of Degree 2 or less and with width of attached gingiva for which the existing Guided Tissue Regeneration (GTR) and bone graft implantation treatment are considered appropriate
4. Those for whom supportive periodontal treatment is applicable (the tooth has the potential to be maintain for at least 3 years), in accordance with usual post-operative procedures following flap operation and GTR treatment
5. Those whose oral hygiene is well established and who are able to perform appropriate tooth brushing and cleaning following instructions of the investigators and/or sub-investigators after investigational drug administration
6. Those 18-years-old and <65-years-old Those who has at least one tooth (e.g. wisdom tooth) that is need to be extracted and the patient agrees the tooth extraction.
7. Those who understand the purposes of the trial and are capable of making an independent decision to comply with trial requirements
8. Those who are able to visit our hospital in accordance with the trial schedule

Exclusion Criteria:

1. Those administered a calcium antagonist during the 4 weeks preceding the surgery
2. Those in need of administration of adrenal cortical steroid (equivalent to>20 mg/day of Predonin) within 4 weeks after the surgery
3. Those scheduled to undergo a surgical operation in the vicinity of the tooth to investigate within 36 weeks after surgery
4. Those with coexisting mental or consciousness disorder
5. Those with coexisting malignant tumour or history of the same
6. Those with coexisting diabetes (HbA1C >6.5%)
7. Those in an extremely poor nutritional condition (serum albumin concentration <2 g/dL)
8. Those with 200 mL of blood drawn during the 4 weeks preceding the surgery
9. Those administered another investigational drug during the 24 h preceding investigational drug administration
10. Those with coexisting disorder of the kidney, liver, blood and/or circulatory system (Grade 2 or above)
11. Those who are either pregnant, possibly pregnant or breast-feeding, or who hope to become pregnant during the period of the trial
12. Those with a previous history of hypersensitivity to any biological active drugs
13. Those who smoke more than 10 pieces of cigarettes
14. Those who are involved in the research team of this trial
15. Others who the investigators or sub-investigators determined as unsuitable for the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Periodontal bone regeneration | 1 year
  The main outcome measures in the study protocol were: rate of increase in alveolar bone height and millimeter of clinical attachement level (CAL) regained. In addition, we examined whether and to what extent adverse events, for which causal relationships with the use of PDL cell were not ruled out, emerged. We set rate of increase in alveolar bone height as the most statistically important outcome (primary outcome).

SECONDARY OUTCOMES:
Clinical parameters | 3 months -12 months
  pocket depth (PD), attachment level (AL), and tooth mobility (TM)

CONTACTS AND LOCATIONS:
Overall Officials: Songtao Shi, Ph.D., Study Director — School of Stomatology, Fourth Military Medical Univeristy; Ostrow School of Dentistry, University of Southern California
Locations (1):
- School of Stomatology, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Chen FM, Jin Y. Periodontal tissue engineering and regeneration: current approaches and expanding opportunities. Tissue Eng Part B Rev. 2010 Apr;16(2):219-55. doi: 10.1089/ten.TEB.2009.0562. PMID 19860551
- [Background] Sonoyama W, Liu Y, Fang D, Yamaza T, Seo BM, Zhang C, Liu H, Gronthos S, Wang CY, Wang S, Shi S. Mesenchymal stem cell-mediated functional tooth regeneration in swine. PLoS One. 2006 Dec 20;1(1):e79. doi: 10.1371/journal.pone.0000079. PMID 17183711
- [Background] Seo BM, Miura M, Gronthos S, Bartold PM, Batouli S, Brahim J, Young M, Robey PG, Wang CY, Shi S. Investigation of multipotent postnatal stem cells from human periodontal ligament. Lancet. 2004 Jul 10-16;364(9429):149-55. doi: 10.1016/S0140-6736(04)16627-0. PMID 15246727
- [Background] Feng F, Akiyama K, Liu Y, Yamaza T, Wang TM, Chen JH, Wang BB, Huang GT, Wang S, Shi S. Utility of PDL progenitors for in vivo tissue regeneration: a report of 3 cases. Oral Dis. 2010 Jan;16(1):20-8. doi: 10.1111/j.1601-0825.2009.01593.x. PMID 20355278
- [Background] Liu Y, Zheng Y, Ding G, Fang D, Zhang C, Bartold PM, Gronthos S, Shi S, Wang S. Periodontal ligament stem cell-mediated treatment for periodontitis in miniature swine. Stem Cells. 2008 Apr;26(4):1065-73. doi: 10.1634/stemcells.2007-0734. Epub 2008 Jan 31. PMID 18238856
- [Background] Fang D, Seo BM, Liu Y, Sonoyama W, Yamaza T, Zhang C, Wang S, Shi S. Transplantation of mesenchymal stem cells is an optimal approach for plastic surgery. Stem Cells. 2007 Apr;25(4):1021-8. doi: 10.1634/stemcells.2006-0576. Epub 2006 Dec 14. PMID 17170063
- [Background] Park JC, Kim JM, Jung IH, Kim JC, Choi SH, Cho KS, Kim CS. Isolation and characterization of human periodontal ligament (PDL) stem cells (PDLSCs) from the inflamed PDL tissue: in vitro and in vivo evaluations. J Clin Periodontol. 2011 Aug;38(8):721-31. doi: 10.1111/j.1600-051X.2011.01716.x. Epub 2011 Mar 30. PMID 21449989
- [Background] Krasner P, Verlander P. Stem cells in dentistry and medicine: the dentist's role. Dent Today. 2011 Jan;30(1):128, 130-4; quiz 135. PMID 21306072
- [Background] Simsek SB, Keles GC, Baris S, Cetinkaya BO. Comparison of mesenchymal stem cells and autogenous cortical bone graft in the treatment of class II furcation defects in dogs. Clin Oral Investig. 2012 Feb;16(1):251-8. doi: 10.1007/s00784-010-0486-7. Epub 2010 Nov 18. PMID 21086003
- [Background] Yang Y, Rossi FM, Putnins EE. Periodontal regeneration using engineered bone marrow mesenchymal stromal cells. Biomaterials. 2010 Nov;31(33):8574-82. doi: 10.1016/j.biomaterials.2010.06.026. Epub 2010 Sep 15. PMID 20832109
- [Background] Washio K, Iwata T, Mizutani M, Ando T, Yamato M, Okano T, Ishikawa I. Assessment of cell sheets derived from human periodontal ligament cells: a pre-clinical study. Cell Tissue Res. 2010 Sep;341(3):397-404. doi: 10.1007/s00441-010-1009-1. Epub 2010 Jul 15. PMID 20632035
- [Background] Iwata T, Yamato M, Zhang Z, Mukobata S, Washio K, Ando T, Feijen J, Okano T, Ishikawa I. Validation of human periodontal ligament-derived cells as a reliable source for cytotherapeutic use. J Clin Periodontol. 2010 Dec;37(12):1088-99. doi: 10.1111/j.1600-051X.2010.01597.x. PMID 20618549
- [Background] Yang ZH, Jin F, Zhang XJ, Liu X, Zhang YF, Liu JQ, Duan YZ, Jin Y. A novel possible strategy based on self-assembly approach to achieve complete periodontal regeneration. Artif Organs. 2010 Jul;34(7):603-9. doi: 10.1111/j.1525-1594.2009.00991.x. Epub 2010 Jun 10. PMID 20545657
- [Background] Wei N, Gong P, Liao D, Yang X, Li X, Liu Y, Yuan Q, Tan Z. Auto-transplanted mesenchymal stromal cell fate in periodontal tissue of beagle dogs. Cytotherapy. 2010 Jul;12(4):514-21. doi: 10.3109/14653241003709702. PMID 20370352
- [Derived] Chen FM, Gao LN, Tian BM, Zhang XY, Zhang YJ, Dong GY, Lu H, Chu Q, Xu J, Yu Y, Wu RX, Yin Y, Shi S, Jin Y. Treatment of periodontal intrabony defects using autologous periodontal ligament stem cells: a randomized clinical trial. Stem Cell Res Ther. 2016 Feb 19;7:33. doi: 10.1186/s13287-016-0288-1. PMID 26895633